CLINICAL TRIAL: NCT06899737
Title: Monitoring and Outreach for Maternal Safety Postpartum
Acronym: MOMSPostpartum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KDH Research & Communication (Industry)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025-02-03; 1R43MD019206-01 (NIH)
Record Dates: First submitted 2025-03-20; First posted 2025-03-28 (Actual); Results first posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Postpartum; Women; Community Health Workers; Knowledge; High-risk; Self Efficacy; Intention; Attitude
Keywords: Community health workers; Postpartum; Support for high risk postpartum women; Women
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Intervention Model Description: Community health workers will be randomly assigned to either the treatment group, which will complete the MOMS Postpartum course, or the control group, which will not receive the training during the study period. Both groups will complete pretest and posttest assessments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment: MOMS Postpartum course (Experimental): Community health workers (CHWs) in the treatment group will complete the MOMS Postpartum course online training program. They will engage with the training materials, apply learned concepts, and complete pretest and posttest assessments to measure changes in their knowledge, skills, attitudes, intentions and self-efficacy.
  Interventions: Other: MOMS Postpartum Course
- Control (No Intervention): Community health workers (CHWs) in the control group will not receive access to the MOMS Postpartum course training during the study period. Their will continue their usual work without the additional training while also completing pretest and posttest assessments to allow for comparison with the treatment group.

INTERVENTIONS:
Other: MOMS Postpartum Course — Online professional development training for CHWs on outreach and support for high-risk postpartum mothers
  Arms: Treatment: MOMS Postpartum course

SUMMARY:
Two arm study, intervention and control, to explore the impact of an online training program to help community health workers (CHWs) conduct effective outreach to support postpartum mothers, particularly those at higher risk for complications.

DETAILED DESCRIPTION:
The investigators will use a randomized, two-group, pretest/posttest design to test the efficacy of the MOMS Postpartum course and explore the following research question: To what extent does exposure to the MOMS Postpartum course increase CHWs' knowledge, skills, attitudes/beliefs, self-efficacy, and intentions to provide support to postpartum mothers?

MOMS Postpartum course is set in context of imperative need of assisting postpartum mothers in the U.S. and working with CHWs after pregnancy to have better maternal outcomes, particularly among high-risk mothers. Researchers worked with subject matter experts, CHWs, and the intended audience to ensure the MOMS Postpartum course reflects the specific needs of postpartum mothers; minimize counter-productive duplications of services and resource expenditure; and create empowered opportunities for CHWs to conduct outreach with high-risk postpartum mothers. MOMS Postpartum course will provide an effective, low-cost, evidence-based, professional development curriculum to train CHWs to provide support to postpartum mothers and fill a gap in care.

The Principal Investigator (PI), with input from the subject matter experts and CHWs, developed necessary research materials, including the recruitment protocols, evaluation instrumentation, and human subjects consent materials . The PI also outlined the appropriate statistical analysis methods. All procedure documents were reviewed by the KDHRC Institutional Review Board before the evaluation launch.

Investigators will recruit participants through evaluation partners who will disseminate the study information to CHWs via electronic notifications and flyers. Evaluation partners include CHW Association of Rochester, Center for Health Innovation, and other CHW organizations. The notifications and flyers provide information about the goal of the study, participant eligibility, and a link to an eligibility form. Once a potential participant completes the eligibility form and s/he is eligible for the study, they will receive a link to a consent form located on a secure online platform.

After consent and enrollment into the study, CHWs will complete a pretest survey and be randomly assigned to the intervention or control group. The intervention group will be exposed to MOMS Postpartum course and will complete an online posttest survey after completing the online modules. The control group participants will not be exposed to the MOMS Postpartum course and will complete a posttest one week after completing the pretest. Participant responses to pretest and posttest survey measures will be linked using non-personal identifiers.

The investigators will download and export the data from Alchemer into an encrypted Excel file and import the raw data into STATA. The investigators will match the pretest and posttest responses using the random assigned identifiers and conduct analyses to test for the effect of MOMS Postpartum course exposure on changes in CHWs' knowledge, skills, attitudes/beliefs, perceived self-efficacy, and intentions to conduct outreach to postpartum mothers.

The initial feasibility criterion is: Statistically significant (p<0.05) and positive relationship between exposure to MOMS Postpartum course and increased knowledge among the intervention group in comparison to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 18 years old.
* Must self-identify as a community health worker (CHW).
* Must live in the United States.
* Must have six months of field experience. KDHRC defines "field experience" as conducting outreach activities in their community, for example, working with clients in a clinic, conducting home visits, or educating clients at health fairs or community events.
* Must be an active CHW. KDHRC defines "active" as conducting outreach activities, such as working with clients in a clinic, conducting home visits, or educating clients at health fairs or community events, in the last six months.
* Must have Internet access either at home or at work to access the lessons and/or online surveys.

Exclusion Criteria:

* None

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2025-03-05 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dexter L Cooper, MPH, Principal Investigator — KDH Research & Communication
Locations (1):
- KDH Research & Communication, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment: MOMS Postpartum Course | Control
Started | 60 | 60
Completed | 41 | 53
Not Completed | 19 | 7
Not completed — Lost to Follow-up | 19 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment: MOMS Postpartum Course | Control | Total
Number analyzed (Participants) | 41 | 53 | 94
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.61 (13.70) | 44.73 (11.12) | 43.79 (12.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 50 | 88
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 15 | 23
  Not Hispanic or Latino | 33 | 37 | 70
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 30 | 32 | 62
  White | 5 | 7 | 12
  More than one race | 1 | 4 | 5
  Unknown or Not Reported | 5 | 8 | 13
Years of CHW experience [Mean (Standard Deviation); unit: years] | 4.41 (3.51) | 6.70 (7.23) | 5.70 (5.99)
Highest education [Number; unit: participants]
  High school diploma/GED | 5 | 6 | 11
  Some college, no degree | 13 | 15 | 28
  Bachelor's degree or higher | 15 | 25 | 40
  Other | 7 | 7 | 14
  Prefer not to answe | 1 | 0 | 1
Hours of CHW training in the last 12 months [Count of Participants; unit: Participants]
  0-5 hours | 9 | 4 | 13
  6-10 hours | 3 | 5 | 8
  11-20 hours | 2 | 8 | 10
  21-29 hours | 5 | 5 | 10
  30+ hours | 22 | 30 | 52
  Not reported | 0 | 1 | 1
CHW certification [Count of Participants; unit: Participants]
  State recognized certification | 30 | 31 | 61
  None | 8 | 16 | 24
  Not sure | 3 | 6 | 9
Volunteer or paid position [Count of Participants; unit: Participants]
  Paid | 26 | 34 | 60
  Volunteer | 5 | 11 | 16
  Both paid and volunteer | 10 | 8 | 18

OUTCOME MEASURES:

1. Primary Outcome: Knowledge Pretest Score
Description: Multiple-choice questions on content related to postpartum care, self-care practices, and needs of postpartum mothers based on information from the MOMS Postpartum course lessons. The score is reported on a scale of 0 to 100, calculated as the percentage of correctly answered questions. Higher scores indicate greater knowledge.
Time Frame: Pretest (Baseline)
Population: One participant excluded for missing data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment: MOMS Postpartum Course | Control
Number analyzed (Participants) | 40 | 53
score on a scale | 77.08 (13.31) | 80.19 (11.23)
Statistical Analysis 1: Comparison: Treatment: MOMS Postpartum Course vs Control; Test type: Superiority; p = 0.32, t-test, 2 sided; Mean Difference (Final Values) = -2.55, 95% CI 2-sided [-7.64 to 2.55], Standard Error of Mean 2.56

2. Primary Outcome: Knowledge Posttest Score
Description: as for outcome 1
Time Frame: Posttest (1 week after baseline)
Population: One participant excluded for missing data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment: MOMS Postpartum Course | Control
Number analyzed (Participants) | 40 | 53
score on a scale | 85.63 (11.16) | 79.56 (13.53)
Statistical Analysis 1: Comparison: Treatment: MOMS Postpartum Course vs Control; Test type: Superiority; p = 0.18, t-test, 2 sided; Mean Difference (Final Values) = 4.18, 95% CI 2-sided [-1.94 to 10.30], Standard Error of Mean 3.08

3. Primary Outcome: Skills Pretest Score
Description: Likert scale ranging from 1 (no experience) to 10 (extensive experience), with a higher score being a better outcome, on conducting education and outreach to postpartum mothers and how to support postpartum mothers
Time Frame: Pretest (Baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment: MOMS Postpartum Course | Control
Number analyzed (Participants) | 41 | 53
score on a scale | 6.64 (2.69) | 6.52 (2.43)
Statistical Analysis 1: Comparison: Treatment: MOMS Postpartum Course vs Control; Test type: Superiority; p = 0.71, t-test, 2 sided; Mean Difference (Final Values) = 0.18, 95% CI 2-sided [-0.81 to 1.18], Standard Error of Mean 0.50

4. Primary Outcome: Skills Posttest Score
Description: as for outcome 3
Time Frame: Posttest (1 week after baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment: MOMS Postpartum Course | Control
Number analyzed (Participants) | 41 | 53
score on a scale | 8.23 (1.26) | 7.77 (2.11)
Statistical Analysis 1: Comparison: Treatment: MOMS Postpartum Course vs Control; Test type: Superiority; p = 0.32, t-test, 2 sided; Mean Difference (Final Values) = 0.61, 95% CI 2-sided [-0.03 to 1.24], Standard Error of Mean 0.32

5. Primary Outcome: Self-efficacy Pretest Score
Description: Likert scale ranging from 1 (strongly disagree) to 10 (strongly agree) to measure CHWs' beliefs that they can effectively support postpartum mothers
Time Frame: Pretest (Baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment: MOMS Postpartum Course | Control
Number analyzed (Participants) | 41 | 53
score on a scale | 7.94 (2.15) | 7.89 (0.36)
Statistical Analysis 1: Comparison: Treatment: MOMS Postpartum Course vs Control; Test type: Superiority; p = 0.91, t-test, 2 sided; Median Difference (Final Values) = 0.05, 95% CI 2-sided [-0.82 to 0.92], Standard Error of Mean 0.44

6. Primary Outcome: Self-efficacy Posttest Score
Description: Likert scale ranging from 1 (no experience) to 10 (extensive experience), with a higher score being a better outcome, to measure CHWs' beliefs that they can effectively support postpartum mothers
Time Frame: Posttest (1 week after baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment: MOMS Postpartum Course | Control
Number analyzed (Participants) | 41 | 53
score on a scale | 8.81 (1.13) | 8.12 (2.11)
Statistical Analysis 1: Comparison: Treatment: MOMS Postpartum Course vs Control; Test type: Superiority; p = 0.059, t-test, 2 sided; Median Difference (Final Values) = 0.69, 95% CI 2-sided [-0.03 to 1.42]

7. Primary Outcome: Attitudes Pretest Score
Description: Likert scale ranging from 1 (strongly disagree) to 10 (strongly agree) on attitudes conducting education and outreach to postpartum mothers and how to support postpartum mothers
Time Frame: Pretest (Baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment: MOMS Postpartum Course | Control
Number analyzed (Participants) | 41 | 53
score on a scale | 8.20 (0.32) | 8.31 (0.26)
Statistical Analysis 1: Comparison: Treatment: MOMS Postpartum Course vs Control; Test type: Superiority; p = 0.79, t-test, 2 sided; Median Difference (Final Values) = -0.10, 95% CI 2-sided [-0.92 to 0.71], Standard Error of Mean 0.41

8. Primary Outcome: Attitudes Posttest Score
Description: as for outcome 7
Time Frame: Posttest (1 week after baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment: MOMS Postpartum Course | Control
Number analyzed (Participants) | 41 | 53
score on a scale | 8.99 (0.16) | 8.50 (0.26)
Statistical Analysis 1: Comparison: Treatment: MOMS Postpartum Course vs Control; Test type: Superiority; p = 0.14, t-test, 2 sided; Mean Difference (Final Values) = 0.50, 95% CI 2-sided [-0.16 to 1.15], Standard Error of Mean 0.33

9. Primary Outcome: Intentions Pretest Score
Description: Likert scale ranging from 1 (extremely unlikely) to 10 (extremely likely) on intentions conducting education and outreach to postpartum mothers and how to support postpartum mothers
Time Frame: Pretest (Baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment: MOMS Postpartum Course | Control
Number analyzed (Participants) | 41 | 53
score on a scale | 8.02 (2.23) | 8.36 (1.90)
Statistical Analysis 1: Comparison: Treatment: MOMS Postpartum Course vs Control; Test type: Superiority; p = 0.42, t-test, 2 sided; Mean Difference (Final Values) = -0.34, 95% CI 2-sided [-1.19 to 0.50], Standard Error of Mean 0.43

10. Primary Outcome: Intentions Posttest Score
Description: as for outcome 9
Time Frame: Posttest (1 week after baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment: MOMS Postpartum Course | Control
Number analyzed (Participants) | 41 | 53
score on a scale | 8.69 (1.43) | 8.36 (1.90)
Statistical Analysis 1: Comparison: Treatment: MOMS Postpartum Course vs Control; Test type: Superiority; p = 0.37, t-test, 2 sided; Mean Difference (Final Values) = 0.33, 95% CI 2-sided [-0.40 to 1.07], Standard Error of Mean 0.37

11. Secondary Outcome: Satisfaction at Posttest
Description: Likert scale ranging from 1 (strongly disagree) to 10 (strongly agree), with a higher score being a better outcome, to measure CHWs' satisfaction with the course, interactive experiences, and offline resources and measure the extent to which CHWs would recommend the course
Time Frame: Posttest (1 weeks after baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment: MOMS Postpartum Course
Number analyzed (Participants) | 41
score on a scale | 9.12 (1.00)

12. Other Pre Specified Outcome: Change in Knowledge Scores From Pretest to Posttest
Description: At both pretest and posttest, we asked all participants the same multiple choice knowledge questions on content related to postpartum care, self-care practices, and needs of postpartum mothers based on information from the MOMS Postpartum course lessons, which we will average to create a composite knowledge score for each participant ranging from 0 to 100. A score of 0 meant a participant got zero questions correct while a score of 100 meant a participant got all questions correct. We will average these composite scores across all participants for both groups to create mean scores. We then subtracted pretest scores from posttest scores and will average these changes for all participants. Positive scores mean a gain in knowledge and a higher scores mean higher gains from baseline to posttest.
Time Frame: From pretest to posttest (1 week)
Population: One participant excluded for missing data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment: MOMS Postpartum Course | Control
Number analyzed (Participants) | 40 | 53
score on a scale | 6.09 (20.58) | -0.63 (12.32)
Statistical Analysis 1: Comparison: Treatment: MOMS Postpartum Course vs Control; Test type: Superiority; p = 0.05, t-test, 2 sided; Mean Difference (Final Values) = 6.72, 95% CI 2-sided [-0.06 to 13.51], Standard Error of Mean 3.42

13. Other Pre Specified Outcome: Change in Skills Scores From Pretest to Posttest
Description: Likert scale ranging from 1 (no experience) to 10 (extensive experience), with a higher score being a better outcome, on conducting education and outreach to postpartum mothers and how to support postpartum mothers. We will average ratings from each question to create an average composite rating for each participant, then average these composite scores for both groups. We will then subtract pretest scores from posttest scores and averaged these changes for all participants. Positive scores mean a gain in skills and higher scores mean higher gains from baseline to posttest.
Time Frame: From pretest to posttest (1 week)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment: MOMS Postpartum Course | Control
Number analyzed (Participants) | 41 | 53
score on a scale | 1.71 (1.96) | 1.17 (1.36)
Statistical Analysis 1: Comparison: Treatment: MOMS Postpartum Course vs Control; Test type: Superiority; p = 0.23, t-test, 2 sided; Mean Difference (Final Values) = 0.42, 95% CI 2-sided [-0.26 to 1.11], Standard Error of Mean 0.35

14. Other Pre Specified Outcome: Change in Self-Efficacy Scores From Pretest to Posttest
Description: Likert scale ranging from 1 (strongly disagree) to 10 (strongly agree), with a higher score being a better outcome, on conducting education and outreach to postpartum mothers and how to support postpartum women. We will average ratings from each question to create an average composite rating for each participant, then average these composite scores for both groups. We will then subtract pretest scores from posttest scores and average these changes for all participants. Positive scores mean a gain in self-efficacy and higher scores mean higher gains from baseline to posttest.
Time Frame: From pretest to posttest (1 week)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment: MOMS Postpartum Course | Control
Number analyzed (Participants) | 41 | 53
score on a scale | 0.87 (1.83) | 0.23 (1.79)
Statistical Analysis 1: Comparison: Treatment: MOMS Postpartum Course vs Control; Test type: Superiority; p = 0.08, t-test, 2 sided; Mean Difference (Final Values) = 0.65, 95% CI 2-sided [-0.09 to 1.39], Standard Error of Mean 0.37

15. Other Pre Specified Outcome: Change in Attitudes Scores From Pretest to Posttest
Description: Likert scale ranging from 1 (strongly disagree) to 10 (strongly agree) on attitudes conducting education and outreach to postpartum mothers and how to support postpartum mothers. We will average ratings from each question to create an average composite rating for each participant, then average these composite scores for both groups. We will then subtract pretest scores from posttest scores and averaged these changes for all participants. Positive scores mean a gain in attitudes and higher scores mean higher gains from baseline to posttest.
Time Frame: From pretest to posttest (1 week)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment: MOMS Postpartum Course | Control
Number analyzed (Participants) | 41 | 53
score on a scale | 0.79 (1.68) | 0.19 (1.90)
Statistical Analysis 1: Comparison: Treatment: MOMS Postpartum Course vs Control; Test type: Superiority; p = 0.11, t-test, 2 sided; Mean Difference (Final Values) = 0.59, 95% CI 2-sided [-0.15 to 1.35], Standard Error of Mean 0.38

16. Other Pre Specified Outcome: Change in Intention Scores From Pretest to Posttest
Description: Likert scale ranging from 1 (extremely unlikely) to 10 (extremely likely) on intentions conducting education and outreach to postpartum mothers and how to support postpartum mothers. We averaged ratings from each question to create an average composite rating for each participant, then averaged these composite scores for both groups. We then subtracted pretest scores from posttest scores and averaged these changes for all participants. Positive scores mean a gain in intentions and higher scores mean higher gains from baseline to posttest.
Time Frame: From pretest to posttest (1 week)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment: MOMS Postpartum Course | Control
Number analyzed (Participants) | 41 | 53
score on a scale | 0.67 (1.79) | 0.00000008 (1.53)
Statistical Analysis 1: Comparison: Treatment: MOMS Postpartum Course vs Control; Test type: Superiority; p = 0.05, t-test, 2 sided; Mean Difference (Final Values) = 0.67, 95% CI 2-sided [-0.01 to 1.36], Standard Error of Mean 0.34

ADVERSE EVENTS:
Time Frame: **not collected**
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Treatment: MOMS Postpartum Course | Control
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-02-03): https://cdn.clinicaltrials.gov/large-docs/37/NCT06899737/Prot_SAP_000.pdf